CLINICAL TRIAL: NCT07355452
Title: Comparing Outcomes Of Single Layer Versus Multilayer Leg Closure Techniques Following Great Saphenous Vein Harvesting For CABG
Acronym: CABG
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Cardiovascular Diseases, Pakistan (Other)
Responsible Party: Principal Investigator, Dr khuzaima Tariq, Assistant Professor and program Director (cardiac surgery training), National Institute of Cardiovascular Diseases, Pakistan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-54/2025; no funding/grants (Other: No funding/grants)
Record Dates: First submitted 2025-12-01; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Surgical Wound Infection; Hematoma; Seroma Following Procedure; Prolonged Hospital Stay; Readmission Rates; Asepsis Score; Surgical Site Infection (SSI)
Keywords: SSI; single vs multilayer wound closure; ASEPSIS SCORE; CABG; GSV harvesting
MeSH Terms: conditions — Surgical Wound Infection; Hematoma

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multi-layer Closure(MLC) (Active Comparator): Multi-layer Closure: multi-layer closure after great saphenous vein harvesting for CABG
  Interventions: Procedure: Multi-layer closure (MLC)
- Single-layer Closure(SLC) (Experimental): Single-layer Closure: single-layer closure after great saphenous vein harvesting for CABG
  Interventions: Procedure: singlelayer closure for leg wound

INTERVENTIONS:
Procedure: Multi-layer closure (MLC) — Coronary artery bypass grafting remains a cornerstone in the management of coronary artery disease, with frequent use of the great saphenous vein as a conduit. While surgical techniques for vein harvesting have evolved, the optimal closure method for the resulting incision remains controversial . The technique employed for closure after vein harvesting can vary, with single-layer and multi-layer closure techniques . Multi-layer closure has remained a standard approach providing adequate tissue approximation and wound healing . However, in recent years, single-layer closure with suction drainage has emerged as a potential alternative, with proponents suggesting it may lead to improved wound healing, reduced complications, and enhanced patient outcomes
  Arms: Multi-layer Closure(MLC)
Procedure: singlelayer closure for leg wound — Multilayer closure for leg wound
  Arms: Single-layer Closure(SLC)

SUMMARY:
This study aims to address the knowledge gap by comparing the outcomes of single-layer and multi-layer leg closure techniques following great saphenous vein harvesting for Coronary artery bypass grafting.

Research question:

1. Does single-layer closure compared to multi-layer closure result in better postoperative outcomes in patients undergoing great saphenous vein harvesting for CABG
2. To evaluate the incidence of postoperative complications (e.g., infection, hematoma, wound dehiscence, seroma) associated with single-layer vs. multi-layer closure techniques.

participants will follow in OPD after 1 week , their wounds will be examined and assessment will be recorded.

DETAILED DESCRIPTION:
This study aims to address the knowledge gap by comparing the outcomes of single-layer and multi-layer leg closure techniques following great saphenous vein harvesting for Coronary artery bypass grafting.

Research question:

1. Does single-layer closure compared to multi-layer closure result in better postoperative outcomes in patients undergoing great saphenous vein harvesting for CABG
2. To evaluate the incidence of postoperative complications (e.g., infection, hematoma, wound dehiscence, seroma) associated with single-layer vs. multi-layer closure techniques.

participants will follow in OPD after 1 week , their wounds will be examined and assessment will be recorded.

Primary Endpoints: ASEPSIS SCORE Secondary Endpoints: Length of hospital stay, infection, hematoma, wound dehiscence, seroma Follow-up at 2 weeks. Readmission for leg wound complications or interventions

ELIGIBILITY:
Sample Selection Sampling Technique: Non-probability consecutive sampling

Inclusion Criteria:

* elective CABG
* Both male and female patients
* Patient of age between 18-70 years
* Patients of consenting surgeons will be included in the study after elaboration of study protocol

Exclusion Criteria:

* Patients with previous leg surgery,
* peripheral vascular disease,
* obesity, BMI; >30kg/m 2 .(weight in kilogram, height in meters)
* varicose veins
* those undergoing total arterial revascularization
* emergency CABG

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-06-30 (Actual); Primary Completion 2026-02-25 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of postoperative leg wound complications (e.g., infection, hematoma, wound dehiscence, seroma) associated with single-layer vs. multi-layer closure techniques | 7 days
  Number of patients enrolled in each group will be assessed for incidence of postoperative complications (e.g., infection, hematoma, wound dehiscence, seroma) associated with single-layer vs multilayer closure techniques using ASEPSIS score. Primary outcomes noticed in both arms will be compared within first 7 days postoperatively. A validated tool called ASEPSIS score will be used and score will be calculated for all patients registered in this study.
Incidence of postoperative leg wound complications (e.g., infection, hematoma, wound dehiscence, seroma, re-suturing, readmission) associated with single-layer vs. multi-layer closure techniques | 14 days
  Number of patients enrolled in each group will be assessed for incidence of postoperative complications (e.g., infection, hematoma, wound dehiscence, seroma) associated with single-layer vs multilayer closure techniques using ASEPSIS score. Primary outcomes noticed in both arms will be compared within first 7 days postoperatively. A validated tool called ASEPSIS score will be used and score will be calculated for all patients registered in this study.

CONTACTS AND LOCATIONS:
Overall Officials: Khuzaima Tariq, Principal Investigator — National Institute of Cardiovascular Diseases
Locations (1):
- National Institute of cardiovascular diseases, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided